CLINICAL TRIAL: NCT05004948
Title: Resistance Exercise Versus Aerobic Exercise Combined With Metformin Therapy in the Treatment of Type 2 Diabetes: A 12-Week Comparative Clinical Study
Brief Title: Exercise Intervention Combined With Metformin in the Treatment of Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prince Sattam Bin Abdulaziz University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RHPT/018/029
Record Dates: First submitted 2021-08-07; First posted 2021-08-13 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Type 2 Diabetes
Keywords: Resistance exercise; Aerobic exercise; Metformin; Insulin resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Resistance exercise group (Active Comparator): This group has conducted a resistance exercise program (50-60% of 1RM, for 40-50 min) thrice weekly for consecutive twelve weeks plus metformin medication.
  Interventions: Other: Exercise training
- Aerobic exercise program (Active Comparator): This group has conducted an aerobic exercise program ( 50-70% maxHR, for 40-50 min) thrice weekly for consecutive twelve weeks plus metformin medication.
  Interventions: Other: Exercise training
- Metformin group (No Intervention): This group received only metformin without any exercise intervention.

INTERVENTIONS:
Other: Exercise training — The first group conducted a resistance exercise program (REP, 50-60% of 1RM, for 40-50 min) combined with metformin, the second group conducted an aerobic exercise program (AEP, 50-70% maxHR, for 40-50 min) combined with metformin, and the third group received only metformin without exercise intervention (Met group). The study program was conducted thrice weekly for consecutive twelve weeks.
  Other Names: Resistance and aerobic exercise program
  Arms: Aerobic exercise program; Resistance exercise group

SUMMARY:
Background: Both exercise and metformin are used to control blood glucose levels in patients with type 2 diabetes mellitus (T2DM), while no previous studies have investigated the effect of resistance exercise combined with metformin versus aerobic exercise with metformin in T2DM patients. This study was conducted to compare the effects of resistance exercise combined with metformin versus aerobic exercise with metformin in T2DM patients.

DETAILED DESCRIPTION:
Background: Both exercise and metformin are used to control blood glucose levels in patients with type 2 diabetes mellitus (T2DM), while no previous studies have investigated the effect of resistance exercise combined with metformin versus aerobic exercise with metformin in T2DM patients. This study was conducted to compare the effects of resistance exercise combined with metformin versus aerobic exercise with metformin in T2DM patients.

Methods: A total of fifty-seven T2DM patients with a mean age of 46.2±8.3 years were randomized to three study groups; each group included nineteen patients. The first group conducted a resistance exercise program (REP, 50-60% of 1RM, for 40-50 min) combined with metformin, the second group conducted an aerobic exercise program (AEP, 50-70% maxHR, for 40-50 min) combined with metformin, and the third group received only metformin without exercise intervention (Met group). The study program was conducted thrice weekly for consecutive twelve weeks. Fasting blood glucose (FBG), glycated hemoglobin (HbA1c), homeostatic model assessment of insulin resistance (HOMA-IR), and maximal oxygen uptake (VO2max) were evaluated before and after study intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of T2DM
* Glycated hemoglobin (HbA1c) ≥8.0%
* A previous inactive lifestyle
* Not receiving insulin or diabetic medications except for metformin
* Metformin dosage of 1000-1500 mg daily.

Exclusion Criteria:

* Cancer
* Pregnancy
* Corticosteroid medications
* Uncontrolled systemic diseases
* Any physical limits that affect exercise training

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Change in Glycated hemoglobin% (HbA1c%) | Pre and post 12-week intervention
  It was were evaluated before and after study intervention by collecting blood samples after fasting 10-12 hours overnight.

SECONDARY OUTCOMES:
Fasting blood glucose (FBG) | Pre and post 12-week intervention
  It was were evaluated before and after study intervention by collecting blood samples after fasting 10 hours overnight.
homeostatic model assessment of insulin resistance (HOMA-IR) | Pre and post 12-week intervention
  It was were evaluated before and after study intervention by collecting blood samples after fasting 10-12 hours overnight.
The maximum oxygen uptake (VO2max) | Pre and post 12-week intervention
  It was assessed pre- and post-intervention on an electrical cycle ergometer (PravoMedics, Salt Lake City, UT, USA) based on an incremental cycling exercise test. The protocol was initiated with 2 min warming-up at a workload of 30W followed every 2 min by a 30W increase until the patient reaches volitional exhaustion.
  During exercise protocol, the oxygen consumption was measured using a breath-by-breath gas analyzer device (FitMate Cosmed, Rome, Italy). VO2max was estimated as the highest average value of 30-s. The technician encouraged the individuals during the last part of the test to generate the maximal effort until voluntary termination. 5-10 min after ending the incremental phase, VO2max value was verified through conducting a supramaximal constant effort to exhaustion based on the criteria for determining VO2max.

CONTACTS AND LOCATIONS:
Overall Officials: Walid Kamal Abdelbasset, PhD, Principal Investigator — Prince Sattam Bin Abdulaziz University
Locations (1):
- Prince Sattam bin Abdulaziz University, Al Kharj, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No